CLINICAL TRIAL: NCT05954390
Title: The Effect of LentinexHP® on Quality of Life in Stage IV Colorectal Cancer: a Randomized, Parallel-group, Placebo-controlled Study
Brief Title: The Effect of LentinexHP® on Quality of Life in Stage IV Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GlycaNova AS (Industry)
Collaborators: OPIS USA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNAS-22-01
Record Dates: First submitted 2023-05-31; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-05

CONDITIONS: Change in Mood; Change in Personality
Keywords: B-Glucan; Quality-of-Life; Colerectal Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded, randomized study. Only the administering pharmacist will have access to the randomization tables
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Therapy (Active Comparator): The active comparator intervention is a solution containing undenatured beta-glucans
  Interventions: Dietary Supplement: Undenatured beta-glucan solution
- Placebo (Placebo Comparator): The placebo comparator intervention is the same solution used in the active comparator intervention except it does not contain any beta-glucans
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Undenatured beta-glucan solution — The active comparator is a solution containing undenatured beta-glucans
  Arms: Active Therapy
Other: Placebo — The placebo comparator is the same solution as the active therapy except it does not contain any undenatured beta-glucans
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind parallel-group, placebo-controlled study. that will last 40 weeks and will focus on Quality of Life.36 Subjects with stage IV metastatic colorectal cancer will be referred for study inclusion. Patients will be randomly assigned (1:1 ratio) to take 2 ml of LentinexHP or placebo orally twice a day (a total of 6 mg). Products will be dispensed to allow administration of the product for six weeks. Each bottle of LentinexHP or placebo contains 30 mL, which at 1.5 mg/mL will provide dosage for approximately five days. The patients will periodically complete the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Quality of Life (QoL) instrument, the short form 36 (SF-36), the Fatigue Symptom Inventory (FSI), and the QoL questionnaire used in the previous LentinexHP QoL study.

DETAILED DESCRIPTION:
This is a randomized, double-blind parallel-group, placebo-controlled study. Subjects with stage IV metastatic colorectal cancer identified by the Principal Investigator or other qualified oncologists will be referred for potential study inclusion.

* Baseline Visit (Week 1) After written informed consent and verification of eligibility criteria, patients will be randomly assigned (1:1 ratio) to take 2 ml of LentinexHP or placebo orally twice a day (a total of 6 mg). Products will be dispensed to allow administration of the product for six weeks. Each bottle of LentinexHP or placebo contains 30 mL, which at 1.5 mg/mL will provide dosage for approximately five days.

Patient demographics, blood chemistries, complete blood count (CBC), and vital signs, will be obtained from the patient's medical records and included as part of the study.

The patients will then complete the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Quality of Life (QoL) instrument, the short form 36 (SF-36), the Fatigue Symptom Inventory (FSI), and the QoL questionnaire used in the previous LentinexHP QoL s

* Visit 2 (Week 6) After six weeks, patients will be asked to return to the clinic and return used/unused bottles of LentinexHP or placebo for compliance evaluation. Patients will evaluate their QoL over the first six weeks of supplementation through the FACT-C, SF-36, FSI and the QoL questionnaire used in a prior LentinexHP study assessing QoL. Any self-perceived adverse events (AE) will be discussed with the patient. The Investigator will also review cancer treatments, vital signs and blood data (if available) to assess for any changes that might have occurred over the first six-week period.
* Visit 3 (Week 12) Patients will return to the clinic with their used/unused bottles of LentinexHP or placebo and again fill out the various QoL questionnaires. As in Visit 2, cancer treatments, blood data and vital signs obtained from medical records will be reviewed.

At this time patients will be given the option of taking LentinexHP free of charge for an additional 40 weeks. If they select that option, the sponsor will send them a 6-week supply of LentinexHP along with the four questionnaires to complete. After receiving the completed questionnaires for each 6-week period, another shipment of LentinexHP for the next 6 weeks will automatically be sent to the patients. Patients will be called every six weeks to enquire about survival, cancer treatments and any adverse events.

The duration of the study for each patient is 12 weeks, extending up to one year for patients opting to continue supplementation after the initial 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age 18 years or older.
* Male or female.
* Patients with stage IV metastatic colorectal cancer with less than three metastatic sites.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Patients starting on 1st or 2nd line chemotherapy with a 5-fluorouracil (5-FU) based regimen with or without biologics.

Exclusion Criteria:

* Patients with known or suspected hypersensitivity to any of the components of the test food supplement.
* Pregnant or breastfeeding.
* Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization (COVID-19 drugs recommended by local regulatory authorities are permitted).
* Patients who in the opinion of the treating physician should not participate in this program.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: * The primary objective of the study is to explore the effect of LentinexHP versus placebo as an add-on non-drug therapy to improve QoL in patients with stage IVmetastatic colorectal cancer. | 12 Weeks
  The primary Instrument to be used for evaluation of the QoL is a validated 27-item questionnaire (FACT-C) designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The FACT-C questionnaire assess the quality of life concerns pertinent to colorectal cancer patients.at weeks, 0 (baseline), 6 and 12. The scale has a numerical value from 0 to 9, where the rating of 0 means the patient feels worse than they did at a previous time point, and a rating of 9 means the patient feels much better than they did at a previous time point. Values between 0 and 9 reflect relative feelings on that day.

SECONDARY OUTCOMES:
Secondary Objective (Outcome 2)* A secondary objective of this study is to evaluate the patients' self-perception of their overall health. | 12 Weeks
  A secondary Instrument to be used for evaluation of the QoL is the validated 36-Item Short Form Survey (SF-36). This is an outcome measure instrument that is often used self-reported measure of health. SF-36 scores range from 0 (worst) to 100 (best) (5). This instrument addresses health concepts from the patient's perspective. The SF-36 questionnaire assesses the quality of life at weeks 0 (baseline), 6 and 12.

OTHER OUTCOMES:
Secondary Objective (Outcome 3)* An additional secondary objective of this study is to evaluate the level of fatigue experienced by the patients during the study | 12 Weeks
  The Fatigue Symptom Inventory (FSI), is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life since the last test period. FSI Severity is measured with four items using an 11-point scale (0 = Not at all fatigued to 10 = As fatigued as I could be). The FSI questionnaire assesses fatigue at weeks 0 (baseline), 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Stoil Borchev, MD, Principal Investigator — CLINECA EAD Hospital, Medical Oncology
Locations (1):
- CLINECA EAD Hospital, Haskovo, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
All data will be available to other researchers and/or recognized organizations upon request, at the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available for an extended period of time (i.e. 5 years) upon completion of the study
Access Criteria: All qualified researchers and government institutions will be able to obtain the data